CLINICAL TRIAL: NCT04689945
Title: Metabolomic Profiling of Erector Spinae Plane Block for Breast Cancer Surgery
Brief Title: Metabolomic Profiling of Erector Spinae Plane Block* for Breast Cancer Surgery
Acronym: ESP
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hazal Ekin GÜRAN AYTUĞ. MD, Anesthesiology Resident, MD, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2020-12/898
Record Dates: First submitted 2020-11-19; First posted 2020-12-30 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: erector spinae plane block; breast cancer; anesthesia and cancer; nerve block and cancer; cancer prognosis
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Morphine; Analgesics, Opioid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Morphine: 30 patients who received intravenous morphine intraoperatively, without regional block application
  Interventions: Drug: Morphine
- Erector Spinae Block: 30 patients who had preoperative esp block but did not use morphine during or after surgery
  Interventions: Procedure: Erector Spinae Block
- Control: 30 patients who received multimodal analgesia methods other than ESP block or IV morphine
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Morphine — PREOPERATIVE ANALGESIA: None
  INTRAOPERATİVE ANALGESIA:
  1. Paracetamol 1000 mg IV
  2. Morphine 0,1 mg/kg IV
  POSTOPERATIVE ANALGESIA IV Morphine Patient-Controlled Analgesia (PCA) Rescue analgesic: IV paracetamol
  Other Names: Opioid
  Groups: Morphine
Procedure: Erector Spinae Block — PREOPERATIVE ANALGESIA:
  Ultrasonography (USG) guided ESP block:T4 spinal level, %0,25 concentration 20 ml, single injection
  INTRAOPERATİVE ANALGESIA:
  1. Paracetamol 1000 mg IV
  2. dexketoprofen 50 mg IV
  POSTOPERATIVE ANALGESIA IV PCA with tramadol Rescue analgesic: IV paracetamol
  Other Names: Plane block
  Groups: Erector Spinae Block
Drug: Control — PREOPERATIVE ANALGESIA: none
  INTRAOPERATİVE ANALGESIA:
  1. Paracetamol 1000 mg IV
  2. Dexketoprofen 50 mg IV
  POSTOPERATIVE ANALGESIA IV PCA with tramadol Rescue analgesic: IV paracetamol
  Other Names: other
  Groups: Control

SUMMARY:
Worldwide, breast cancer is the most common cancer among women, and its incidence and mortality rates are expected to increase significantly in the next years. It remains a major health problem. There is a vast area on breast cancer and immunity that still needs to be researched. Do anesthetic techniques and medication preferences effect immune responses? If so how they effect breast cancer outcomes is unclear.

On this trial, the investigators are searching anesthetic techniques affect on inflammatory and immune responses.

DETAILED DESCRIPTION:
Breast cancer is the most frequently encountered surgery among all cancer surgeries. Although it is a well known procedure for anesthesiologists, it is still unclear whether anesthesiology effects immune responses. Cancer therapies often use immune therapies such as Bevacizumab (a monoclonal antibody which targets Vascular Endothelial Growth Factor), Trastuzumab(a monoclonal antibody for Herceptin (HER2/Neu) mutation) how anesthetics effect VEGF stays unclear.

Opioids are commonly used to provide analgesia for cancer pain, and functional opioid receptors have been identified on natural killer (NK) cells, the lymphocytes responsible for surveillance and elimination of cancer cells.[4] Anesthesiologists have well founded concerns about using morphine during cancer surgeries.

Regional anesthetic techniques commonly used on cancer surgeries.The activation of sensory neurons during pain enhances tumor progression and metastatic potential. Regional anesthesia blocks somatic nociception and inhibits sympathetic preganglionic outflow (functional sympathectomy) during surgery. Moreover regional anesthesia, by blocking sympathetic nervous system output, induces a prevalence of parasympathetic tone. Local anesthetics can also modulate autonomic receptors. For these reasons, more studies are needed to investigate the action of regional anesthetic neuromodulation on cancer progression.[11]

The Erector Spinae Plane Block (ESP block) is most often performed on thoracic paraspinal levels, causes sympathetic blockage. Sympathetic block has been studied on central neuraxial blocks but the sympathetic block caused by the ESP block and immune responses remain unclear.

Sympathetic block inhibits hyperbolic immune responses after surgery, therefore enhances postoperative rate of acceleration on cytokine levels. The investigators propose that ESP block improves immune responses and improved immune responses have better clinical outcomes for patients with breast cancer. Improved immune responses decrease length of stay (LOS), enhance postoperative recovery, analgesia and quality of life. Therefore allows better patient experience about procedures.

The investigators will take 90 patients who will undergo a breast cancer operation and compare vitals (heart rate, blood pressure, oxygen saturation), Numeric Rating Scales (NRS), Vascular Endothelial Growth Factor (VEGF) responses, systemic immune inflammatory indexes, cortisol levels, CRP and Procalcitonin levels between three groups; opioid analgesia group(group M), ESP block group(group E), non-opioid non-ESP group (group P).

The investigators' main focus is immune alterations after anesthesia techniques. Anesthesiologist keep track of pain scores after surgery. this trials secondary outcome focuses on pain management after surgery.

ELIGIBILITY:
Inclusion criteria:

1. Should be female
2. Should be between 18-65 years old
3. Diagnosed with unilateral primary breast cancer
4. Are decided to have mastectomy surgery
5. Stage 1-2 breast cancer (T0-1-2, N0-1, M0)

Exclusion criteria from the:

1. Being allergic to the anesthetics
2. Previously had breast operation other than diagnostic biopsy
3. Presence of a malignancy history on the other breast
4. Diagnosed with Inflammatory breast cancer
5. Having a risk score of The American Society of Anaesthesiologists (ASA) risk score 3 and above
6. Contraindications for regional block(Allergies for local anesthetics, Anatomic application difficulties, Coagulopathies)
7. Hormone usage
8. NRS score greater than 3 before the operation
9. Opioid or steroid usage before the operation
10. Rheumatologic history
11. Sickness or drug usage that might cause immunosuppression
12. Chemotherapy and/or radiotherapy history
13. Concomitant history of previous malignancy
14. History of Coronary Artery Disease, Peripheral Vascular Disease that may affect VEGF
15. Chronic smoking
16. Chronic obstructive pulmonary disease
17. Presence of infection at the time of surgery
18. Hypothalamus, Pituitary, adrenal gland dysfunction
19. Autoimmune diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will evaluate unilateral breast cancer patients from Ankara Dr. Abdurrahman Yurtaslan Oncology Train and Research Hospital who will undergo Mastectomy procedure.
  The investigators will exclude patients who no longer want to participate at any part of the trial.
  A total of 90 patients' data will be collected.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Metabolomic profiling of ESP block for breast cancer surgery | 24 hours postoperatively
  Metabolomic profiling of 3 groups will be performed with liquid chromatography mass spectrometrt (LCMS) and Quadrupole time-of-flight (Q-TOF).

SECONDARY OUTCOMES:
Defining the change in preoperative (baseline), postoperative hour 24 Vascular Endothelial Growth Factor (VEGF) levels between the morphine group (group M), the ESP block group (group E), and the control group (group c). | change from baseline VEGF at 24 hours postoperatively
  The investigators will measure VEGF preoperative(baseline), postoperative hour 24 from blood analysis.
  Normal ranges of serum VEGF were 62-707 pg/ml.
Defining the change in preoperative (baseline), postoperative hour 1, postoperative hour 24 cortisol levels between the morphine group (group M), the ESP block group (group E), and the control group (group c). | change from baseline cortisol up to 24 hours postoperatively
  The investigators will measure cortisol preoperative(baseline),postoperative hour 1, postoperative hour 24 from blood analysis.
  Serum cortisol normal range for adults 8 am to 4pm: 5-25 mcg/dL
Defining the change in preoperative (baseline), postoperative hour 1, postoperative hour 24 C-reactive Protein levels between the morphine group (group M), the ESP block group (group E), and the control group (group c). | change from baseline CRP up to 24 hours postoperatively
  The investigators will measure CRP preoperative(baseline), postoperative hour 1, postoperative hour 24 from blood analysis.
  CRP normal reading is less than 10mg/L.
Defining analgesic effects between the morphine group (group M), the ESP block group (group E), and the control group (group c) on patients who had breast cancer surgery. | End of surgery up to 24 hours postoperatively
  The investigators will evaluate patients' pain score with numeric rating scale (NRS) postoperative hour 1, 2, 12, 24 and compare NRS between the control group (group c), the ESP block group (group E) and intravenous morphine group (group M)
  The investigators will compare NRS between two groups at postoperative hour 1, 2, 12, 24.
  The most common form of NRS is a horizontal line with an eleven point numeric range, from 0 (patient with no pain) to 10 (patient with the worst pain possible).
Tramadol consumption between the ESP block group and the control group | End of surgery up to 24 hours postoperatively
  The investigators will record total opioid consumption via Patient-Controlled Analgesia devices.

CONTACTS AND LOCATIONS:
Overall Officials: hazal ekin güran aytug, resident, Principal Investigator — Dr. Abdurrahman Yurtaslan Oncology Train and Research Hospital
Locations (1):
- Dr.Abdurrahman Yurtaslan Ankara Oncology Train and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available starting 6 months from publication.
Access Criteria: IPD will be shared with other clinical experimenters in order to serve as an example to similar studies and to demonstrate the reliability of the study. Consent forms of the participants, preoperative evaluation and postoperative follow-up forms, blood results evaluating inflammatory responses, postoperative analgesia need follow-up form will be open to sharing.

REFERENCES:
- [Background] Harbeck N, Gnant M. Breast cancer. Lancet. 2017 Mar 18;389(10074):1134-1150. doi: 10.1016/S0140-6736(16)31891-8. Epub 2016 Nov 17. PMID 27865536
- [Background] Bates JP, Derakhshandeh R, Jones L, Webb TJ. Mechanisms of immune evasion in breast cancer. BMC Cancer. 2018 May 11;18(1):556. doi: 10.1186/s12885-018-4441-3. PMID 29751789
- [Background] Sen Y, Xiyang H, Yu H. Effect of thoracic paraspinal block-propofol intravenous general anesthesia on VEGF and TGF-beta in patients receiving radical resection of lung cancer. Medicine (Baltimore). 2019 Nov;98(47):e18088. doi: 10.1097/MD.0000000000018088. PMID 31764844
- [Background] Maher DP, Walia D, Heller NM. Morphine decreases the function of primary human natural killer cells by both TLR4 and opioid receptor signaling. Brain Behav Immun. 2020 Jan;83:298-302. doi: 10.1016/j.bbi.2019.10.011. Epub 2019 Oct 15. PMID 31626971
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Demirci U, Yaman M, Buyukberber S, Coskun U, Baykara M, Uslu K, Ozet A, Benekli M, Bagriacik EU. Prognostic importance of markers for inflammation, angiogenesis and apoptosis in high grade glial tumors during temozolomide and radiotherapy. Int Immunopharmacol. 2012 Dec;14(4):546-9. doi: 10.1016/j.intimp.2012.08.007. Epub 2012 Aug 29. PMID 22940539
- [Background] Sultan SS. Paravertebral block can attenuate cytokine response when it replaces general anesthesia for cancer breast surgeries. Saudi J Anaesth. 2013 Oct;7(4):373-7. doi: 10.4103/1658-354X.121043. PMID 24348286
- [Background] Deegan CA, Murray D, Doran P, Moriarty DC, Sessler DI, Mascha E, Kavanagh BP, Buggy DJ. Anesthetic technique and the cytokine and matrix metalloproteinase response to primary breast cancer surgery. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):490-5. doi: 10.1097/AAP.0b013e3181ef4d05. PMID 20975461
- [Background] Sen S, Koyyalamudi V, Smith DD, Weis RA, Molloy M, Spence AL, Kaye AJ, Labrie-Brown CC, Morgan Hall O, Cornett EM, Kaye AD. The role of regional anesthesia in the propagation of cancer: A comprehensive review. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):507-522. doi: 10.1016/j.bpa.2019.07.004. Epub 2019 Jul 31. PMID 31791567
- [Background] Forget P, Aguirre JA, Bencic I, Borgeat A, Cama A, Condron C, Eintrei C, Eroles P, Gupta A, Hales TG, Ionescu D, Johnson M, Kabata P, Kirac I, Ma D, Mokini Z, Guerrero Orriach JL, Retsky M, Sandrucci S, Siekmann W, Stefancic L, Votta-Vellis G, Connolly C, Buggy D. How Anesthetic, Analgesic and Other Non-Surgical Techniques During Cancer Surgery Might Affect Postoperative Oncologic Outcomes: A Summary of Current State of Evidence. Cancers (Basel). 2019 Apr 28;11(5):592. doi: 10.3390/cancers11050592. PMID 31035321